CLINICAL TRIAL: NCT04092699
Title: Cone Beam Computed Tomographic Segmentation in Volumetric Measurements of Maxillary Sinus Using Different Soft Wares: A Validity and Reliability Study
Brief Title: CBCT Segmentation in Volumetric Measurements of MS Using Different Soft Wares: A Validity and Reliability Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ashraf Hussien, principle investigator, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Dentistry
Record Dates: First submitted 2019-09-11; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Sinus Volume; CBCT Segmentation
Keywords: CBCT; maxillary sinus; segmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Other): CBCT Dicom file of patient has been scanned will be used for measurements of maxillary sinus volume by different software
  Interventions: Device: semiautomatic software
- skulls (Other): CBCT Dicom file of patient has been scanned will be used for measurements of maxillary sinus volume by different software
  Interventions: Device: semiautomatic software

INTERVENTIONS:
Device: semiautomatic software — semiautomatic segmentation is as accurate as the direct volume of maxillary sinus and as well as the manual segmentation.
  Other Names: Mimics medical 19.; Romexis; On Demand 3D

SUMMARY:
Cone Beam Computed Tomography (CBCT) has been used to assess the volume of the maxillary sinus using the manual and semi-automatic segmentation. The majority of researches stressed on the reduced accuracy of the automatic segmentation when compared to the real volume. Regarding the semi-automatic segmentation, there are researches assessed the volumetric measurement of the maxillary sinus and they reported that there is no significant difference between semi- automatic and the manual segmentation in CT.

DETAILED DESCRIPTION:
Automatic segmentation is believed to be less time consuming and more accurate in assessment of structures with regular border but fairly assessed the structures with irregular border like paranasal sinuses. The semi-automatic software is efficient and accurate as manual tracing with significant reduction in inter-observer variability and time . On the other hand, all neighboring contacting voxels located within a defined range (threshold) of similar HU values of different adjacent tissues may be measured so over calculation or under calculation could be suspected

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria of participants of the In vitro part of the study:

* Skulls with intact walls of maxillary sinus.
* Skulls with dentulous or edentulous jaws.

Exclusion criteria of participants:

* Skulls with missing parts of the maxilla that could be caused from traumatic injuries, diseases and space occupying lesions of maxilla.
* Skulls with severe mutilation caused by environmental decay.

Inclusion Criteria of participants of the In vivo part of the study:

* Patients without any pathosis affects maxillary sinus.
* Patients with dentulous or edentulous jaws.

Exclusion criteria of participants:

* Patients with traumatic injuries, diseases and space occupying lesions of maxilla.
* Patients with sinus lifting or surgeries.
* Patients with mucosal thickening more than 3mm

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of CBCT semiautomatic segmentation in Volumetric measurements of maxillary sinus. | 1 year
  validity and reliability

CONTACTS AND LOCATIONS:
Overall Officials: Reham Ashraf, master, Principal Investigator — Reham Ashraf Hussien

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berberi A, Bouserhal L, Nader N, Assaf RB, Nassif NB, Bouserhal J, Salameh Z. Evaluation of Three-Dimensional Volumetric Changes After Sinus Floor Augmentation with Mineralized Cortical Bone Allograft. J Maxillofac Oral Surg. 2015 Sep;14(3):624-9. doi: 10.1007/s12663-014-0736-3. Epub 2014 Dec 24. PMID 26225054
- [Result] Alsufyani NA, Flores-Mir C, Major PW. Three-dimensional segmentation of the upper airway using cone beam CT: a systematic review. Dentomaxillofac Radiol. 2012 May;41(4):276-84. doi: 10.1259/dmfr/79433138. PMID 22517995
- [Result] El H, Palomo JM. Measuring the airway in 3 dimensions: a reliability and accuracy study. Am J Orthod Dentofacial Orthop. 2010 Apr;137(4 Suppl):S50.e1-9; discussion S50-2. doi: 10.1016/j.ajodo.2010.01.014. PMID 20381759